CLINICAL TRIAL: NCT03483428
Title: Adaptation and Pilot Implementation of the Family Check-Up for Deaf and Hard of Hearing Children
Brief Title: Adaptation and Pilot Testing of a Behavioral Parent Training Program for Parents of Deaf and Hard of Hearing Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Responsible Party: Principal Investigator, Christina Studts, Assistant Professor, University of Kentucky
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-0460-F6A
Record Dates: First submitted 2018-03-23; First posted 2018-03-30 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Hearing Loss; Behavior Disorders; Parenting
MeSH Terms: conditions — Hearing Loss; Mental Disorders | interventions — Organization and Administration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parent Coaches (Experimental): Parent coaches will complete interventionist training and supervision in the "Family Check-Up," an evidence-based behavioral parent training (BPT) program, including in the adaptations for families with DHH children. Each parent coach will deliver the intervention to 5 parent-child dyads.
  Interventions: Behavioral: Interventionist training and supervision
- Parent-Child Dyads (Experimental): Parents and children will receive the adapted "Family Check-Up" behavioral parent training (BPT) intervention delivered by parent coaches.
  Interventions: Behavioral: Behavioral parent training

INTERVENTIONS:
Behavioral: Interventionist training and supervision — Online and in-person training and weekly supervision with licensed clinical social worker while delivering the "Family Check-Up" to 5 families.
  Arms: Parent Coaches
Behavioral: Behavioral parent training — Up to 6 sessions of the "Family Check-Up" program, involving discussions, assessments, feedback, and skills training with a parent coach.
  Arms: Parent-Child Dyads

SUMMARY:
Despite being more likely than typical hearing children to experience disruptive behavior problems, children who are deaf and hard of hearing (DHH) rarely receive behavioral interventions to prevent the long-term costly outcomes of behavior problems. This pilot project will systematically adapt an evidence-based behavioral parent training (BPT) intervention to increase its acceptability and relevance for parents of young DHH children. Two parents of DHH children will be trained in the adapted BPT for DHH children. They will each deliver the intervention to five families with DHH preschool-aged children.

ELIGIBILITY:
Parent/Caregivers and Children:

Inclusion Criteria:

* Parent/caregiver is age 18 years or older
* Parent/caregiver is the custodial guardian of a deaf or hard of hearing (DHH) child
* DHH child is 2-5 years old
* DHH child has used hearing aid(s) and/or cochlear implant(s) for > 6 months
* Parent/caregiver is able to read English and either speak/understand English or use American Sign Language

Exclusion Criteria:

* Active child protective services case
* DHH child of interest has been diagnosed with a severe developmental delay, severe autism, debilitating neurological condition, etc.
* Parent/caregiver has already accessed behavioral health services for the DHH child

Parent Coaches/Interventionists:

Inclusion Criteria:

* Age 18 years or older
* Parent of a DHH child
* Able to speak, understand, and read English

Exclusion Criteria:

- None

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2018-04-11 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Feasibility: Enrollment | 2 weeks after final parent-child dyad completes the study
  Proportion of parents agreeing to enroll in the intervention out of all parents approached

SECONDARY OUTCOMES:
Feasibility: Number of sessions completed | 2 weeks after final parent-child dyad completes the study
  Number of sessions completed by each enrolled parent
Interventionist fidelity | 2 weeks after final parent-child dyad completes the study
  Fidelity ratings of two recorded sessions per interventionist
Feasibility: usability of battery of measures | 2 weeks after final parent-child dyad completes the study
  Proportion of missing data across and within instruments for parent, child, and interventionist outcome measures
Acceptability: parent satisfaction | 10 weeks after parent baseline
  European Parent Satisfaction Scale about Early Intervention (EPASSEI) - adapted; range: 20 (high satisfaction) to 100 (low satisfaction)
Acceptability: interventionist satisfaction | 2 weeks after final parent-child dyad completes the study
  Therapist Satisfaction Index (TSI)

CONTACTS AND LOCATIONS:
Overall Officials: Christina Studts, PhD, Principal Investigator — University of Kentucky, Dept of Health, Behavior & Society; Matthew Bush, MD, PhD, Principal Investigator — University of Kentucky, Dept of Otolaryngology
Locations (1):
- University of Kentuckyi, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No